CLINICAL TRIAL: NCT04531267
Title: Ratio of Dietary Calcium to Magnesium on Cardiovascular Risk of High-risk Population: an Intervention Study
Brief Title: Ratio of Dietary Calcium to Magnesium on Cardiovascular Risk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2019781H
Record Dates: First submitted 2020-06-16; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-05

CONDITIONS: Hypertension; Nutritional and Metabolic Diseases; Cardiovascular Risk Factor
MeSH Terms: conditions — Hypertension; Nutritional and Metabolic Diseases | interventions — Magnesium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized nutrition (Active Comparator): Participants' diet will be assessed by food frequency questionnaire to obtain calcium and magnesium intake. Individualized dosage of dietary supplements will be provided to maintain a calcium/magnesium ratio as 2.3. Participants will stay with the original medication plan.
  Interventions: Dietary Supplement: Individualized dosage of calcium and magnesium
- Control group (No Intervention): Participants do not receive any supplements, they stay with the original medication plan.

INTERVENTIONS:
Dietary Supplement: Individualized dosage of calcium and magnesium — Participants' diet will be assessed by food frequency questionnaire to obtain calcium and magnesium intake. Individualized dosage of dietary supplements will be provided to maintain a calcium/magnesium ratio as 2.3. Participants will stay with the original medication plan.
  Arms: Individualized nutrition

SUMMARY:
Although the epidemiological studies indicate how magnesium and calcium may interact to affect cardiovascular risk, current clinical trials have not elucidated the associations, particularly among hypertensive patients. To address the research gap, we have to examine how magnesium may influence cardiovascular profile of hypertensive patients via the modification of calcium homeostasis. Meanwhile, large-scale cohorts in China suggested keeping dietary calcium: magnesium ratio within 2.3 can reduce the risk of cardiovascular mortality. The results indicate the potential for individualized nutrition. This study will recruit uncontrolled hypertensive patients taking single drug and investigate whether calcium-magnesium combined supplements help to control their blood pressure. In standardized manner, subjects in the intervention group and the control group (each with 21 subjects) will be assessed for their dietary calcium and magnesium intake in the previous three months, so that researchers can provide calcium and/or magnesium supplements to maintain a calcium/magnesium ratio as 2.3. The effect of supplementation will be evaluated by the blood pressure changes in the 12th week of intervention.

DETAILED DESCRIPTION:
In 2015, the prevalence of hypertension in Chinese adults was 25.2%, which can be translated into 25 million people with hypertension in Guangdong Province. Hypertension is also related to narrowing and occlusion of the cardiovascular vessels. In China, coronary heart disease and stroke are the main causes of death in many provinces, and the early prevention of cardiovascular disease risk in patients with hypertension has become a research direction dedicated to the whole population. Magnesium is the second most abundant intracellular ion in the body, which can regulate vascular tone, and together with calcium leads to changes in vascular smooth muscle tone and contractility. Magnesium deficiency is associated with oxidative stress, inflammation, endothelial dysfunction, platelet aggregation, insulin resistance, and hyperglycemia; in the long run, dietary magnesium deficiency also increases the risk of developing metabolic syndrome, type 2 diabetes, cardiovascular disease, and cancer. However, the impact of nutrients on health is affected by different dietary factors. Calcium and magnesium share different ion receptors or channels, including Calcium-sensing receptor (modulates parathyroid hormone levels, thereby increasing the production of vitamin D), as well as TRPM6 and TRPM7 (modulates the absorption of calcium and magnesium ions). In a large meta-analysis, there is also evidence that calcium supplements may reduce blood pressure in healthy people.

In addition, in epidemiological studies, we can see the interactive relationship between calcium and magnesium. In the American population, when the ratio of calcium to magnesium is <2.8, dietary intake of calcium and magnesium can reduce the risk of colorectal adenoma. However, when the ratio of calcium to magnesium is too low (<2.0), it may also cause adverse effects. According to data from more than 130,000 people in the Shanghai Women's Health Study and the Shanghai Men's Health Study, the median calcium-magnesium ratio (1.7) in the Chinese population is much lower than the calcium-magnesium ratio (3.0) in the US population. When the calcium-magnesium ratio is > 1.7, calcium and magnesium intake can reduce the mortality of cardiovascular disease; but when the calcium-magnesium ratio is <1.7, magnesium intake increases the risk of cardiovascular death in women. Although the interaction between magnesium and calcium can influence cardiovascular risk in epidemiological studies, the current clinical evidence have not fully verified the relationship, especially among hypertensive patients . To substantiate the research findings, it is necessary to explore how calcium-magnesium intervention can improve the cardiovascular risk factors of hypertensive patients. In addition, personalized nutrition intervention is also a research direction to be explored. Unlike the unified dosage in the past, it may be more important to formulate supplements according to individual dietary habits. In 2018, Vanderbilt University's team conducted a clinical trial among 180 healthy adults with personalized magnesium supplements and examined on the effects of blood vitamin D. They adjusted the dose of supplements according to the calcium-magnesium ratio in the diet at baseline to achieve a calcium-magnesium ratio of 2.3, and tested changes in various types of vitamin D in the blood. They found that the effect of magnesium supplements on vitamin D levels varied according to the baseline 25(OH)D concentration. When 25(OH)D levels are higher, magnesium supplements reduced the levels of 25(OH)D3 and 24,25(OH)2D3. But when 25(OH)D is low, magnesium supplements increased the level of 25(OH)D3. This is the first study to use baseline dietary intakes for personalized nutrition interventions, but they have not explored whether interventions can affect cardiovascular risk factors in hypertensive patients. More randomized trials are needed to verify the efficacy of intervention, especially in high-risk populations.

To answer the above questions, this study is a randomized trial to ensure that the highest level of evidence is obtained and will recruit hypertensive patients in Guangdong Provincial People's Hospital. The intervention and control group have the same number of people.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients that received only one type of medication.
* Uncontrolled blood pressure: 140mmHg≤SBP≤149mmHg, 90mmHg≤DBP≤99mmHg.
* Able to sign informed consent and come to follow-up session by themselves.

Exclusion Criteria:

* Type 1 or 2 diabetic patients, or taking anti-diabetic drugs.
* Taking two types or above anti-hypertensive drugs
* Alanine transaminase or Aspartate Transaminase exceeding normal limits for 2 times or above.
* Acute myocardial infarction, heart failure or stroke in the last 6 months.
* Suffering from chronic gastrointestinal diseases
* Taking calcium or magnesium supplements in a regular basis (at least once per week) in the previous year
* In pregnancy or breastfeeding period, or planning to be pregnant
* Other serious diseases (e.g. cancer) that are not eligible for participation
* Participating in other studies.

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline systolic and diastolic blood pressure at 3 months | Assessed at baseline and 3-month follow-up
  measured by sphygmomanometer

SECONDARY OUTCOMES:
Changes from baseline concentration of hemoglobin A1c at 3 months | Assessed at baseline and 3-month follow-up
  measured by blood test to obtain biochemistry profile
Changes from baseline concentration of fasting glucose at 3 months | Assessed at baseline and 3-month follow-up
  measured by blood test to obtain biochemistry profile
Changes from baseline concentration of fasting insulin at 3 months | Assessed at baseline and 3-month follow-up
  measured by blood test to obtain biochemistry profile
Changes from baseline concentration of serum calcium and magnesium at 3 months | Assessed at baseline and 3-month follow-up
  measured by blood test to obtain biochemistry profile
Changes from baseline concentration of urinary calcium and magnesium at 3 months | Assessed at baseline and 3-month follow-up
  measured by urinary test to obtain biochemistry profile
Changes from baseline concentration of urinary creatine at 3 months | Assessed at baseline and 3-month follow-up
  measured by urinary test to obtain biochemistry profile